CLINICAL TRIAL: NCT02871128
Title: Evaluation of Natureheme-iron on Iron Absorption Effect and Anti-oxidation Functions- a Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Evaluation of Natureheme-iron on Iron Absorption Effect and Anti-oxidation Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, You-Cheng Shen, School of Health Diet and Industry Managment, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CS14135; MOST 104-2622-E-040-002 -CC2 (Other Grant/Funding Number: Ministry of Science and Technology)
Record Dates: First submitted 2016-08-15; First posted 2016-08-18 (Estimated); Results first posted 2020-08-28 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Anemia
Keywords: Hemoglobin; serum iron; serum ferritin; Hematocrit; antioxidant
MeSH Terms: conditions — Anemia | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Natureheme-iron (Experimental): Subjects receive 2 capsules per day containing either 1000 mg Fe.
  Interventions: Dietary Supplement: Natureheme-iron
- Placebo (Placebo Comparator): Subjects receive 2 capsules per day containing starch placebo of similar appearance.
  Interventions: Dietary Supplement: Placebo
- supplement (Active Comparator): Subjects receive 1 capsule per day containing either 100 mg Fe.
  Interventions: Drug: supplement

INTERVENTIONS:
Dietary Supplement: Natureheme-iron — An 12 week double-blinded randomized parallel study with 4 week follow-up period was performed in mild anemia subjects. Consenting eligible subjects were receive 2 capsules per day containing either 1000 mg Fe of similar appearance for 12 weeks. The subjects were required to visit at baseline, every 6 weeks during the intervention period (6 weeks), and at follow-up 4 weeks after treatment had ended. During each study visit, fasting blood samples were collected and anthropometric measurements were performed. Compliance was evaluated using a food diary and monitored with biweekly telephone calls.
  Arms: Natureheme-iron
Dietary Supplement: Placebo — An 12 week double-blinded randomized parallel study with 4 week follow-up period was performed in mild anemia subjects. Consenting eligible subjects were receive 2 capsules per day containing either 1000 mg starch placebo of similar appearance for 12 weeks. The subjects were required to visit at baseline, every 6 weeks during the intervention period (6 weeks), and at follow-up 4 weeks after treatment had ended. During each study visit, fasting blood samples were collected and anthropometric measurements were performed. Compliance was evaluated using a food diary and monitored with biweekly telephone calls.
  Arms: Placebo
Drug: supplement — An 12 week double-blinded randomized parallel study with 4 week follow-up period was performed in mild anemia subjects. Consenting eligible subjects were receive 1 capsule per day containing either 100 mg Fe of similar appearance for 12 weeks. The subjects were required to visit at baseline, every 6 weeks during the intervention period (6 weeks), and at follow-up 4 weeks after treatment had ended. During each study visit, fasting blood samples were collected and anthropometric measurements were performed. Compliance was evaluated using a food diary and monitored with biweekly telephone calls.
  Other Names: latte
  Arms: supplement

SUMMARY:
Iron deficiency problem has always been in Taiwan. This is a randomized, double-blind trial. Subjects separate to 3 groups, one group (n = 20) take two Natureheme-iron capsules a day for a total of 12 weeks, another group (n = 20) with the same dose of placebo, and the other group (n = 20) is a commercial iron supplement. Investigators assess whether Natureheme-iron can promote iron absorption and antioxidant effects, and compare the effects with commercial iron supplement. When this study is completed, it will increase the value of Natureheme-iron, and can improve health of Taiwanese.

DETAILED DESCRIPTION:
FAO / WHO noted that iron deficiency is still an important nutritional problem. Iron deficiency problem has always been in Taiwan. This study intends to use the products, Natureheme-iron, using blood of pig to concentration, separation and extracted, and then got natural and clean Natureheme-iron. Natureheme-iron is not just a good iron supplement, while also providing an excellent source of natural protein. This is a randomized, double-blind trial, subjects separate to 3 groups, one group (n = 20) take two Natureheme-iron capsules a day for a total of 12 weeks (1000mg Fe / capsule), another group (n = 20) with the same dose of placebo, and the other group (n = 20) is a commercial iron supplement (100mg Fe). Investigators assess whether Natureheme-iron can promote iron absorption and antioxidant effects, and compare the effects with commercial iron supplement. When this study is completed, it will increase the value of Natureheme-iron, and can improve health of Taiwanese.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects were anemia men or women aged over 20 years old with Hb<=12 g/dl.

Exclusion Criteria:

* Subjects were excluded if subjects had a history of major cardiovascular disease, severe liver dysfunction, insulin-dependent diabetes mellitus or stroke. Subjects were also excluded if they routinely consumed alcohol, were pregnant or unable to comprehend study instructions.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-07; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: You-Cheng Mr Shen, Ph.D., Principal Investigator — Chung Shan Medical University

REFERENCES:
- [Background] Shaw NS, Liu YH. Bioavailability of iron from purple laver (Porphyra spp.) estimated in a rat hemoglobin regeneration bioassay. J Agric Food Chem. 2000 May;48(5):1734-7. doi: 10.1021/jf990759y. PMID 10820087

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Natureheme-iron | Placebo | Supplement
Started | 20 | 20 | 16
Completed | 20 | 19 | 15
Not Completed | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Natureheme-iron | Placebo | Supplement | Total
Number analyzed (Participants) | 20 | 20 | 16 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 19 | 15 | 53
  >=65 years | 1 | 1 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.70 (11.90) | 33.37 (14.61) | 43.40 (15.29) | 39.82 (13.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 5
  Male | 18 | 18 | 15 | 51
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Taiwan | 20 | 19 | 15 | 54

OUTCOME MEASURES:

1. Primary Outcome: The Hemoglobin of the Subjects at Baseline and 6 Weeks
Description: The Hb (g/dl) measure at baseline and 6 weeks and compare the value at 6 weeks minus value at baseline.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Natureheme-iron | Placebo | Supplement
Number analyzed (Participants) | 20 | 19 | 15
g/dl | 0.38 (0.95) | 0.29 (0.91) | 0.57 (0.99)

2. Secondary Outcome: The Changes of Serum Ferritin of the Subjects.
Description: values change of serum ferritin (ng/ml) between before to after 6 weeks
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Natureheme-iron | Placebo | Supplement
Number analyzed (Participants) | 20 | 19 | 15
ng/ml | 5.22 (91.7) | -0.37 (43.98) | 11.86 (75.82)

ADVERSE EVENTS:
Arm/Group | Natureheme-iron | Placebo | Supplement
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/15
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No